CLINICAL TRIAL: NCT02185625
Title: Reduction of Adverse Pregnancy Outcomes With a Smartphone Application in Ghana: a Cluster Randomized Trial
Brief Title: Reduction of Adverse Pregnancy Outcomes With a Smartphone Application in Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other); University of Ghana (Other); Maternity Foundation (Unknown); Augustinus Fonden (Other); Lundbeck Foundation (Other); Edith and Godtfred Kirk Christiansen Foundation (Unknown); Aase and Ejnar Danielsens Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AU201407; AU201407 (Other: Aarhus University, Department of Public Health)
Record Dates: First submitted 2014-07-01; First posted 2014-07-09 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2015-07

CONDITIONS: Postpartum Hemorrhage; Delivery, Obstetric; Stillbirth; Infant Mortality; Midwifery
MeSH Terms: conditions — Postpartum Hemorrhage; Stillbirth; Infant Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Safe Delivery smartphone application (Experimental)
  Interventions: Device: Safe Delivery smartphone application
- Control (No Intervention)

INTERVENTIONS:
Device: Safe Delivery smartphone application — The intervention is the use of a smartphone application called Safe Delivery, designed by University of Copenhagen, Denmark and Maternity Foundation Denmark. The application contains animated videos aimed to train midwives in the prevention and management of postpartum hemorrhage and the treatment of neonatal resuscitation. The instructions in the videos are based on WHO recommendations, and the application is designed to be an on-going tool for midwives, so that they can drill themselves in the emergencies of postpartum hemorrhage and neonatal resuscitation.
  Arms: Safe Delivery smartphone application

SUMMARY:
The purpose of this study is to determine whether use of the Safe Delivery smartphone application by midwives can reduce excess blood loss from bleeding, and infant death during childbirth in Ghanaian women. Moreover, it will be investigated whether the Safe Delivery application can increase midwives' knowledge and skills in managing childbirth.

Fifteen hospitals in Greater Accra, Ghana, will be cluster randomized to either use the Safe Delivery application (intervention), or to no intervention (control). In the intervention hospitals, midwives will be educated in the use of Safe Delivery. Pregnant women will be enrolled at delivery and followed until 7 days postpartum. Data collection will begin July 2014 and is expected to be finished by October 2014.

ELIGIBILITY:
Inclusion criteria for Hospitals:

* Located in the region of Greater Accra.
* The hospital should have at least 10 midwives employed.
* The patient flow for each midwife should be at least 10 deliveries per month.
* The annual average number of deliveries should be at least 1,200.

Inclusion criteria for midwives:

* Should have no leave or vacation from June 17th to September 17th 2014.
* Should have a full time employment at the delivery ward (conducting deliveries 100% of the work time).
* Should be willing and available to participate in an information meeting at the hospital where the balloting among eligible midwives will take place.
* Should give an informed consent to participate in the study.
* Should be willing and available to participate in a workshop July 14th 2014 (this is the day of randomization, and intervention midwives will receive smartphone training).
* Should be willing and available to participate in a workshop September 17th 2014 (to complete an end of study questionnaire, the key feature questionnaire, and control midwives will receive smartphones).
* Should be proficient in English to understand the spoken instructions in the animated videos.

Inclusion criteria for women in labor:

* Should be in active labor.
* Should give informed consent to participate in the study.
* Should give birth vaginally.

The women in labor and their newborn children will be the primary observational units.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3773 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Postpartum Hemorrhage. | Measurements 2 hours after delivery.
  Postpartum Hemorrhage is defined as blood loss greater than 500 ml from bleeding associated with childbirth within first 2 hours postpartum.

SECONDARY OUTCOMES:
Blood loss | Measurements 2 hours after delivery.
  Amount of blood loss (ml) from bleeding associated with childbirth within first 2 hours postpartum.
Key feature questionnaire (KFQ). | At baseline and 2 months after randomization.
  The KFQ questionnaire measures midwives' knowledge in relation to 1) active management of the third stage of labour, 2) treatment of postpartum hemorrhage, 3) manual removal of placenta, and 4) neonatal resuscitation. The midwives' performance will be scored by research assistants by use of the KFQ tool.
Objective structured assessment of technical skill (OSATS). | At baseline and 2 months after randomization.
  The OSATS tool measures midwives' skills in relation to 1) active management of the third stage of labour, 2) treatment of postpartum hemorrhage, 3) manual removal of placenta, and 4) neonatal resuscitation. The midwives' performance will be scored by research assistants by use of the OSATS tool.
Fresh stillbirth | At delivery.
  Delivery of a fetus with a birth weight above 1,000 g birth weight who at birth has no signs of life (breathing, crying or movement) with intact skin.
Neonatal mortality 7 days postpartum. | Within 7 days postpartum.
  A baby born alive with a birth weight above 1000 g who dies within 7 days postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Christina MB Nielsen, BSc, MPH, Principal Investigator — Department of Public Health, Aarhus University, Denmark
Locations (15):
- Ghana (15):
  - Achimota Hospital, Accra
  - Ashaiman Polyclinic, Accra
  - Ga South Municipal Hospital, Accra
  - Ga West Municipal Hospital, Accra
  - Keneshi Polyclinic, Accra
  - La General Hospital, Accra
  - Lekma Hospital, Accra
  - Maamobi General Hospital, Accra
  - Madina Polyclinic, Accra
  - Mamprobi Polyclinic, Accra
  - Ridge Hospital, Accra
  - Shai Osu Doku District Hospital, Accra
  - Tema General Hospital, Accra
  - Tema Polyclinic, Accra
  - Usher Poly (James Town Maternity Home), Accra